CLINICAL TRIAL: NCT02958657
Title: Effect of Exercise Training on the Autonomic Nervous System and Its Correlation With Platelet Aggregability in a Post-myocardial Infarction Population
Brief Title: Effect of Exercise on Platelet Reactivity After Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Talia Falcão Dalçóquio, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12163
Record Dates: First submitted 2016-10-30; First posted 2016-11-08 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Platelet Aggregation; Acute Myocardial Infarction; Exercise Training
Keywords: Platelet function; Autonomic Nervous System; Multiplate® (Multiple Electrode Aggregometry - MEA); VerifyNow®
MeSH Terms: interventions — Exercise; Physical Conditioning, Human; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Training (Experimental): Patients randomized to the training group will start the supervised regular training program 01 month after the myocardial infarction, and it will last for three months.
  Interventions: Other: Exercise Training
- Control Group (No Intervention): Patients in the control group will receive general instructions regarding rehabilitation post-acute myocardial infarction and will be followed for four months after the myocardial infarction.

INTERVENTIONS:
Other: Exercise Training — Supervised exercise training program that includes two workouts per week for three months at a rehabilitation unit.
  Other Names: Physical Activity; Physical Training; Rehabilitation
  Arms: Exercise Training

SUMMARY:
This project aims to evaluate, in recent post-acute myocardial infarction (AMI) patients on dual antiplatelet therapy, the impact of regular exercise training on platelet aggregability and the correlation between the level of platelet aggregability and muscle sympathetic nerve activity (MSNA).

DETAILED DESCRIPTION:
1. Introduction:

   Platelet reactivity is closely involved in the pathophysiology of acute coronary syndromes (ACS). However, despite the development of newer and more effective antiplatelet drugs (among other therapeutic interventions), the risk of ischemic events recurrence after an episode of ACS is still high.

   On the other hand, acute and strenuous exercise, a known trigger of ACS, when performed by untrained individuals, leads to sympathetic hyperactivity and increased platelet aggregability. Contrary to these findings, regular supervised exercise training leads to regulation of the autonomic system with consequent decrease in the incidence of ACS, as shown in previous studies. However, the relationship between regular supervised exercise training on platelet activity in patients post-AMI on dual antiplatelet therapy, has not been previously studied and is the main goal of the present project.
2. Objectives:

   This project aims to evaluate, in recent post-AMI patients on dual antiplatelet therapy, the impact of regular exercise training on platelet aggregability, analyzed by VerifyNowP2Y12® test. Secondary exploratory analysis includes: 1) the influence of acute and strenuous exercise on platelet aggregability measured immediately after the two cardiopulmonary exercise testing (CPET) that patients will be submitted; 2) the correlation between the level of platelet aggregability and MSNA in trained and control groups; 3) the influence of exercise training on platelet aggregability measured by Multiplate® adenosine diphosphate (ADP) test and Multiplate® aspirin (ASPI) test; 4) the influence of exercise training on the mean platelet volume (MPV) and platelet count; 5) the influence of exercise training in other laboratorial parameters as lipids, blood glucose and inflammatory activity; 6) finally, the primary endpoint of the study will be evaluated in different prespecified subgroups such as diabetics, elderly, obese and patients with chronic kidney disease.

   2.1. Primary endpoint of the study: Evaluate the influence of regular supervised exercise training for 3 months on platelet aggregability, analyzed by VerifyNowP2Y12® test, in patients with recent AMI utilizing dual antiplatelet therapy.

   2.2. Main secondary analyses:

   A. Evaluate platelet aggregability immediately after acute exercise before and after the exercise training period; for this propose, blood sample will be drawn immediately after the first and second cardiopulmonary exercise testings, in trained and control groups.

   B. Correlate the platelet aggregability level, evaluated by VerifyNowP2Y12®, Multiplate-ADP®, Multiplate-ASPI®, with the level of MSNA.

   2.3. Other exploratory analyses:

   A. Evaluate the primary endpoint of the study utilizing Multiplate-ASPI® and Multiplate-ADP®;

   B. Evaluate the MPV in trained and control groups, and its correlation with platelet aggregability;

   C. Analyze, in trained and control groups, the following parameters:

   Platelet count; LDL-cholesterol; HDL-cholesterol; Triglycerides; Lipid transference for HDL; Fasting glucose; Glycated hemoglobin; C-reactive protein (CRP) ultrasensitive; B-type natriuretic peptide (BNP); Troponin and Creatine Kinase MB-mass peak obtained during hospitalization; Genetic polymorphisms; Heart rate variability and spontaneous baroreflex control.

   D. Analyze the primary endpoint within the following subgroups, taking into account the parameters obtained during hospitalization:

   Sex (male / female); ST segment elevation myocardial infarction (STEMI) or non-STEMI; Basal heart rate (<70 or ≥ 70 bpm); History of arterial hypertension (presence or absence); LDL levels (<100 or ≥ 100 mg/dL); Age ≥65 years and <65 years; Body Mass Index <30 or ≥ 30 kg / m2; Creatinine clearance (MDRD) <60ml / min / m2 or ≥ 60 ml / min / m2; Current or not smoking; History of diabetes (present or absent); HbA1c <6.5 or ≥ 6.5%; GRACE risk score ≥140 and <140; Beta-blocker use.
3. Methodology:

This is a prospective, randomized study. Patients with stable AMI admitted to a Coronary Care Unit, eligible to participate, will be randomized to a supervised exercise training program for three months at a rehabilitation unit or to a control group not formally trained. Patients who agree to participate will be included after the necessary explanations and the signature of the informed consent form.

3.a. Sample size calculation: To perform the sample calculation, previously published data wich showed platelet agreeability average of 32.9 ± 16 P2Y12 reactions units (PRU) in post-AMI patients on ticagrelor was utilizes. For an expected 35% decrease in platelet aggregability at trained group, and taking into account power of 80% and alpha index of 0.05, including 31 patients in each group is required. Admitting a percentage of losses of 40% given the difficulties inherent in the assessment of the sympathetic activity and adherence to the training program, the initial plan contemplates the inclusion of 90 patients in the study.

4. Study design: Prospective study in which eligible patients with uncomplicated AMI admitted to a Coronary Care Unit will be randomized to performing a exercise training program by three months or for an untrained control group, at a 1:1 or 1:2 rate, in order to adjust for more frequent early follow-up interruptions in exercise training group. All patients included after the necessary explanations and after signing the informed consent form. The patients will be submitted to the collection of material for laboratory evaluation including platelet aggregability tests, the assessment of a CPET in 01 and 04 months of the follow-up (end of treatment). The MSNA will be performed at the end of followup.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for spontaneous STEMI or non-STEMI in patients older than 18 years.

Exclusion Criteria:

* Any condition that contraindicate physical activity;
* Regular exercise training practitioners prior to the ischemic event;
* Planned revascularization in the following 4 months;
* Hospitalization for cardiovascular events in the previous 12 months;
* Ventricular dysfunction, defined as left ventricular ejection fraction (LVEF) <45% on echocardiography, evaluated by Simpson's method);f) Killip class III and IV;
* High risk of arrhythmia and/or second and third degree atrioventricular block;
* Diabetes mellitus requiring intravenous insulin therapy during hospitalization;
* Important chronic kidney disease, defined by creatinine clearance<30ml/min/m2 (estimated by MDRD formula);
* Oral anticoagulation;
* Use of NSAIDs and/or dipyridamole;
* Contraindication to dual antiplatelet therapy;
* Serum hemoglobin level <10 g/dL;
* Use of glycoprotein IIB/IIIA inhibitors in the last 48 hours;
* Terminal illness;
* Liver disease or coagulopathy;
* Refusal to engage in an exercise training program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-10-30; Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Platelet aggregability by VerifyNow-P2Y12® | Before the second CPET (04 months pot-AMI)
  To measure in recent post-AMI patients on dual antiplatelet therapy the impact of 03 months of regular exercise training (starting 30 days after the AMI) on platelet aggregability, analyzed by VerifyNow-P2Y12® test.

SECONDARY OUTCOMES:
Platelet aggregability by Multiplate-ADP® | After the first CPET (01 month post-AMI)
  To analyze the influence of acute and strenuous exercise on platelet aggregability analysed by Multiplate-ADP® immediately after the first CPET.
Platelet aggregability by Multiplate-ASPI® | After the first CPET (01 month post-AMI)
  To analyze the influence of acute and strenuous exercise on platelet aggregability analysed by Multiplate-ASPI® immediately after the first CPET.
Platelet aggregability by Multiplate-ADP® | After the second CPET (04 months post-AMI)
  To analyze the influence of strenuous exercise on platelet aggregability measured by MultiplateADP® immediately after the second CPET.
Platelet aggregability by Multiplate-ASPI® | After the second CPET (04 months post-AMI)
  To analyze the influence of strenuous exercise on platelet aggregability measured by MultiplateASPI® immediately after the second CPET.
Sympathetic activity by MSNA | Before the second CPET (04 months post-AMI)
  To analyze the influence of exercise training on MSNA, measured by microneurography directly from the peroneal nerve and expressed by postganglionic muscle sympathetic nerve recordings burst frequency (bursts per minute).

CONTACTS AND LOCATIONS:
Overall Officials: Talia F Dalçóquio, MD, Principal Investigator — Heart Institute (InCor) University of Sao Paulo Medical School
Locations (1):
- Heart Institute of University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dalcoquio TF, Alves Dos Santos M, Silva Alves L, Bittar Brito Arantes F, Ferreira-Santos L, Pinto Brandao Rondon MU, Furtado RHM, Gehlen Ferrari A, Genestreti Rizzo PR, Salsoso R, Franci A, Moreira Baracioli L, de Nazare Nunes Alves MJ, Negrao CE, Nicolau JC. Effects of exercise on platelet reactivity after myocardial infarction: a randomized clinical trial. Platelets. 2023 Dec;34(1):2139821. doi: 10.1080/09537104.2022.2139821. Epub 2022 Nov 14. PMID 36377063